CLINICAL TRIAL: NCT02804269
Title: Molecular and Imaging Studies of Cardiovascular Health and Disease
Acronym: Biobank
Status: Recruiting | Type: Observational
Sponsor: National Heart Centre Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: 2013/605/C
Record Dates: First submitted 2016-05-31; First posted 2016-06-17 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2013-07

CONDITIONS: Healthy; Dilated Cardiomyopathy; Hypertrophic Cardiomyopathy; Ischemic Heart Disease
Keywords: Healthy Volunteer; Dilated cardiomyopathy; Hypertrophic cardiomyopathy; ischemic heart disease; Cardiovascular Magnetic Resonance Imaging
MeSH Terms: conditions — Cardiomyopathy, Dilated; Cardiomyopathy, Hypertrophic; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood and serum.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Healthy Volunteer: Subjects will undergo the following study procedure: Cardiovascular Magnetic Resonance Imaging and fatmass measurement
  Interventions: Other: Cardiovascular Magnetic Resonance; Other: Fatmass measurement
- Dilated Cardiomyopathy: Subjects will undergo the following study procedure: Cardiovascular Magnetic Resonance Imaging and fatmass measurement
  Interventions: Other: Cardiovascular Magnetic Resonance; Other: Fatmass measurement
- Hypertrophic cardiomyopathy: Subjects will undergo the following study procedure: Cardiovascular Magnetic Resonance Imaging and fatmass measurement
  Interventions: Other: Cardiovascular Magnetic Resonance; Other: Fatmass measurement
- Ischemic heart disease with reduced EF: Subjects will undergo the following study procedure: Cardiovascular Magnetic Resonance Imaging and fatmass measurement
  Interventions: Other: Cardiovascular Magnetic Resonance; Other: Fatmass measurement
- Ischemic heart disease with normal EF: Subjects will undergo the following study procedure: Cardiovascular Magnetic Resonance Imaging and fatmass measurement
  Interventions: Other: Cardiovascular Magnetic Resonance; Other: Fatmass measurement

INTERVENTIONS:
Other: Cardiovascular Magnetic Resonance — For the evaluation of heart function and structure of the cardiovascular system.
Other: Fatmass measurement — It utilizes a scale machine to measure the body fat and skeletal muscle percentage

SUMMARY:
Biobank is a program which collects biological samples, health information and imaging data from consented patients and stored them at the core facility. These information would be used to study the molecular, imaging and outcome studies of cardiovascular health and disease.

DETAILED DESCRIPTION:
This program recruits patient from National Heart Centre Singapore and collects their biological sample, health information and imaging data.The donated biospecimens will be stored indefinitely and used for any future research on molecular, imaging and outcome studies of cardiovascular health and disease.The same biological samples and imaging data will be obtained from consented healthy volunteers for comparison.

ELIGIBILITY:
There is no inclusion/exclusion criteria except for the age limit as this is a repository program.

Inclusion Criteria:

•Subject aged ≥ 16 years and ≤ 90 years.

Exclusion Criteria:

•No

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patient will be recruited from primary care clinic and outpatient clinics from the National Heart Centre Singapore. For healthy volunteer, they will be recruited through poster and advertisement.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2013-07; Primary Completion 2033-07 (Estimated); Study Completion 2033-07 (Estimated)

PRIMARY OUTCOMES:
Numbers of genetic variation in genes known to cause inherited cardiac condition and circulating biomarkers which are linked with DNA changes using advanced sequencing and informatics approaches | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Cook, MBBS,PhD, Principal Investigator — National Heart Centre Singapore
Locations (1):
- National Heart Centre Singapore, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No